CLINICAL TRIAL: NCT02653326
Title: Integrative Technological Platforms for Telerehabilitation for Patients With Heart Surgery: A Pilot Randomised Trial
Brief Title: Technological Platforms and Telerehabilitation in Heart Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Valparaiso (Other)
Collaborators: Hospital Dr. Gustavo Fricke (Unknown); Fundación Dr. Jorge Kaplan Meier (Unknown)
Responsible Party: Principal Investigator, Felipe Martinez, Professor, Universidad de Valparaiso
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CEC093-15
Record Dates: First submitted 2016-01-08; First posted 2016-01-12 (Estimated); Results first posted 2019-01-28 (Actual); Last update posted 2019-01-28 (Actual); Status verified 2019-01

CONDITIONS: Cardiovascular Diseases; Cardiac Surgery
Keywords: Tertiary Prevention; Telerehabilitation
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Physical Therapy Modalities; Nutrition Assessment

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Telerehabilitation (Experimental): In addition to routine care, patients in this arm will receive a telerehabilitation strategy comprised by a portable EKG monitor and a smartphone application.
  Interventions: Device: Telerehabilitation Monitors; Procedure: Physical Therapy; Behavioral: Nutritional Counseling; Other: Depression Screening; Drug: Treatment of Comorbidities
- Routine Care (Active Comparator): Patients allocated to routine care will receive care as enforced by current practice guidelines. This care included nutritional counseling, depression screening, drug therapy for the management of comorbidities and physical exercise without telemonitoring.
  Interventions: Procedure: Physical Therapy; Behavioral: Nutritional Counseling; Other: Depression Screening; Drug: Treatment of Comorbidities

INTERVENTIONS:
Device: Telerehabilitation Monitors — After completing a 12-session physical therapy programme and the aforementioned co-interventions, patients will receive a telerehabilitation strategy comprised by electrocardiographic monitoring and a smartphone application aimed at detecting adverse events during exercise activities. These devices will also inform patients and healthcare providers regarding the adequacy of their physical activities in terms of cardiovascular outcomes and the observed changes during treatment.
  Arms: Telerehabilitation
Procedure: Physical Therapy — Physical therapy will be provided in form of twelve 90-minute sessions. Exercises will be tailored to patient needs, but a common goal of reaching an oxygen consumption of 80-90% will be used for every participant.
Behavioral: Nutritional Counseling — Nutritional counseling will be provided in 60-minute group sessions for included participants. A nutritionist will provide education in terms of healthy eating and risk factor modification.
Other: Depression Screening — Participants will be screened for depression using the Hospital Anxiety and Depression scale, which has been validated for Spanish-speaking countries. If depression is confirmed, pharmacologic treatment and/or psychotherapy will be prescribed at the discretion of the attending physician.
Drug: Treatment of Comorbidities — Whenever needed, treatment of comorbid conditions, such as hypertension, diabetes or dyslipidemia, will be provided for study participants.

SUMMARY:
In this randomised, double-blind, pilot study, the investigators aim to assess whether a telerehabilitation strategy could improve outcomes among patients with recent heart surgery. Included participants will receive a comprehensive rehabilitation programme comprised of physical therapy, nutritional counselling, psychological assistance in addition to standard medical care. After 12 sessions of physical therapy, patients will be randomised to receive telerehabilitation with a portable EKG device and a smartphone application or usual care. The primary endpoint for this study is the exercise capacity of included participants, which will be assessed using an ergospirometer at 4 and 8 weeks after randomisation.

DETAILED DESCRIPTION:
As in other Latin-american countries, access to rehabilitation programmes is limited, even though their effectiveness has been proved among patients with heart surgery and endorsed in current practice guidelines. In this randomised trial, the investigators aim to assess whether an integrative technological platform might improve the exercise capacity of patients that have undergone heart surgery.

Eligible patients include adult (>18 years old) patients who have undergone any kind of heart surgery in the Hospital Gustavo Fricke between January and December 2016. Patients will be enrolled within 3 weeks of their cardiac surgery into the trial. Patients with any contraindication to physical exercise (see below), Parkinson's disease, severe dementia or psychiatric comorbidities that preclude the initiation of the programme will be excluded. All patients will receive physical training delivered by a group of physical therapists divided in twelve 90-minute sessions. The overall goal of these sessions will be to obtain a workload of 80% - 90% of maximum oxygen consumption (VO2) as established by ergospirometric assessments (Cardiovit CS-200). In addition to exercise, patients will also receive nutritional support, education, risk factor modification and psychological assessments using the Hospital Anxiety and Depression Scale that has been validated in Spanish-speaking countries.

Randomisation will be performed by a statistician and study personnel will be kept unaware of the specific method used. Patients in the intervention arm will receive a telerehabilitation strategy comprised by a portable EKG device that will be aimed at establishing heart rate, stress responses and recovery times after physical activities. This sensor will be used to monitor compliance with a prescribed physical therapy programme. In addition, a second sensor will be deployed in the form of a smartphone application that will provide alerts for patients and healthcare providers whenever an adverse event is recorded. The application will also provide motivational messages for participants to optimize adherence to the exercise programme, as well as information regarding individual improvements in physical activities.

All patients will undergo an ergospirometry at baseline, 4 weeks and 8 weeks after completion of the initial physical therapy sessions. Clinicians, outcome assessors and analysts well be kept unaware of treatment allocations. All analyses will be undertaken under the intention to treat principle. No prespecified subgroup analyses have been programmed.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (>18 years old)
* Recent cardiac surgery (3 weeks)

Exclusion Criteria:

* Contraindication to physical exercise (unstable angina, acute heart failure, complex ventricular arrythmias, severe (>60mmHg) pulmonary hypertension, endocavitary thrombuses, recent deep venous thrombosis (1 month), severe obstructive cardiomyopathy, symptomatic aortic stenosis, musculoskeletal conditions that make exercise impossible)
* Parkinsons' Disease
* Severe dementia or major psychiatric comorbidities that make adherence or comprehension of the intervention impossible
* Refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-01; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carla Taramasco, Ph.D., Study Director — Universidad de Valparaiso; Felipe T Martinez, M.D., M.Sc, Principal Investigator — Universidad de Valparaiso
Locations (2):
- Chile (2):
  - Fundacion Cardiovascular Dr. Jorge Kaplan Meier, Viña del Mar, Región de Valparaíso
  - Hospital Gustavo Fricke, Viña del Mar, Región de Valparaíso

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Telerehabilitation: In addition to routine care, patients in this arm will receive a telerehabilitation strategy comprised by a portable EKG monitor and a smartphone application. For information regarding the routine care interventions, please see the routine care description from the control group.
  Telerehabilitation Monitors: After completing a 12-session physical therapy programme and the aforementioned co-interventions, patients will receive a telerehabilitation strategy comprised by electrocardiographic monitoring and a smartphone application aimed at detecting adverse events during exercise activities. These devices will also inform patients and healthcare providers regarding the adequacy of their physical activities in terms of cardiovascular outcomes and the observed changes during treatment.
- Routine Care: Patients allocated to routine care will receive care as enforced by current practice guidelines. Specific interventions include:
  Physical Therapy: Physical therapy will be provided in form of twelve 90-minute sessions. Exercises will be tailored to patient needs, but a common goal of reaching an oxygen consumption of 80-90% will be used for every participant.
  Nutritional Counseling: Nutritional counseling will be provided in 60-minute group sessions for included participants. A nutritionist will provide education in terms of healthy eating and risk factor modification.
  Depression Screening: Participants will be screened for depression using the Hospital Anxiety and Depression scale, which has been validated for Spanish-speaking countries. If depression is confirmed, pharmacologic treatment and/or psychotherapy will be prescribed at the discretion of the attending physician.
Period: Overall Study
Arm/Group | Telerehabilitation | Routine Care
Started | 32 | 34
Completed | 22 | 27
Not Completed | 10 | 7
Not completed — Lost to Follow-up | 10 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Telerehabilitation | Routine Care | Total
Number analyzed (Participants) | 32 | 34 | 66
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (11.3) | 60.9 (17.1) | 61.4 (14.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 11 | 22
  Male | 21 | 23 | 44
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 28.2 (3.1) | 26.9 (3.4) | 27.5 (3.3)
Smoker [Count of Participants; unit: Participants] | 24 | 22 | 46
Diabetes mellitus [Count of Participants; unit: Participants] | 11 | 14 | 25
Dyslipidemia [Count of Participants; unit: Participants] | 10 | 12 | 22
Hypertension [Count of Participants; unit: Participants] | 27 | 21 | 48
Sleep apnea [Count of Participants; unit: Participants] | 2 | 0 | 2
Peripheral vascular disease [Count of Participants; unit: Participants] | 2 | 0 | 2
Alcoholism [Count of Participants; unit: Participants] | 5 | 4 | 9
Cancer [Count of Participants; unit: Participants] | 1 | 0 | 1
Chronic obstructive lung disease [Count of Participants; unit: Participants] | 4 | 2 | 6
Heart rate at rest [Mean (Standard Deviation); unit: beats per minute] | 80.9 (13.2) | 83.0 (13.6) | 81.9 (13.3)
Heart rate at anaerobic threshold [Mean (Standard Deviation); unit: beats per minute] | 117.1 (21.8) | 116.4 (18.1) | 116.7 (19.8)
Heart rate during maximum intensity exercises [Mean (Standard Deviation); unit: beats per minute] | 127.0 (23.8) | 126 (22.0) | 126.4 (22.7)
Mechanic load at anaerobic threshold [Mean (Standard Deviation); unit: watts] — The anaerobic threshold is defined as the highest sustained intensity of exercise for which measurement of oxygen uptake can account for the entire energy requirement. The mechanic load at this threshold is usually expressed as watts or Joules/second.
  watts | 62.6 (23.2) | 65.5 (29.6) | 64.1 (26.4)
Mechanic load during maximum intensity exercises [Mean (Standard Deviation); unit: watts] | 80.6 (48) | 81.1 (34.2) | 80.9 (41.4)
Oxygen consumption at rest [Mean (Standard Deviation); unit: mL/Kg/minute] | 0.23 (0.82) | 0.24 (0.80) | 0.23 (0.8)
Oxygen consumption during training [Mean (Standard Deviation); unit: mL/Kg/minute] | 0.84 (0.36) | 0.78 (0.25) | 0.81 (0.30)

OUTCOME MEASURES:

1. Primary Outcome: Exercise Capacity Assessed as Peak Oxygen Consumption at 4 Weeks After Randomisation
Description: Ergospirometric assessment of oxygen consumption (VO2) among study participants.
Time Frame: 4 weeks after randomisation
Population: Ergospirometric evaluations were conducted after the initial physiotherapy phase was completed amongst study participants.
Measure: Mean (Standard Deviation); unit: mL/Kg/minute
Arm/Group | Telerehabilitation | Routine Care
Number analyzed (Participants) | 32 | 34
mL/Kg/minute | 0.92 (0.39) | 0.87 (0.26)
Statistical Analysis 1: Comparison: Telerehabilitation vs Routine Care; Test type: Superiority; p = 0.63, t-test, 2 sided

2. Primary Outcome: Exercise Capacity
Description: Exercise Capacity Assessed as Peak Oxygen Consumption at 8 weeks after randomisation
Time Frame: 8 weeks after randomisation
Population: Outcome assessment after telerehabilitation phase was completed. These are complete-case analyses only. Results using multiple imputation techniques for missing data are given below.
Measure: Mean (Standard Deviation); unit: mL/Kg/minute
Arm/Group | Telerehabilitation | Routine Care
Number analyzed (Participants) | 22 | 27
mL/Kg/minute | 1.0 (0.4) | 0.91 (0.28)
Statistical Analysis 1: Comparison: Telerehabilitation vs Routine Care; Test type: Superiority; p = 0.32, t-test, 2 sided

3. Secondary Outcome: Number of Participants With Adverse Events at 4 Weeks
Description: Development of adverse events during exercise, such as myocardial ischemia or malignant arrhythmias.
Time Frame: 4 weeks after randomisation
Measure: Count of Participants; unit: Participants
Arm/Group | Telerehabilitation | Routine Care
Number analyzed (Participants) | 32 | 34
Participants | 0 | 0

4. Secondary Outcome: Number of Participants With Adverse Events at 8 Weeks
Description: Development of adverse events during exercise, such as myocardial ischemia or malignant arrhythmias.
Time Frame: 8 weeks after randomisation
Measure: Count of Participants; unit: Participants
Arm/Group | Telerehabilitation | Routine Care
Number analyzed (Participants) | 22 | 27
Participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Telerehabilitation | Routine Care
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/34
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/34
Other Adverse Events (participants affected / at risk) | 0/32 | 0/34

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No